CLINICAL TRIAL: NCT07148154
Title: ScreenEC: Development of a Non-invasive IVD for Endometrial Cancer Screening on High-risk Populations
Brief Title: Development of a Non-invasive IVD for Endometrial Cancer Screening on High-risk Populations
Status: Recruiting | Type: Observational
Sponsor: MiMARK Diagnostics, S.L. (Industry)
Collaborators: Hospital Vall d'Hebron (Other)
Responsible Party: Sponsor
Other Study IDs: ScreenEC
Record Dates: First submitted 2025-08-21; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Endometrial Cancer
Keywords: Endometrial Cancer; IVD; In-vitro Diagnostics; Endometrial adenocarcinoma; diagnostics
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Cytological Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — Cytology specimen, cervical sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Consultancy participants: Eligible participants are postmenopausal women presenting with abnormal uterine bleeding (AUB) in a clinical consultation or primary care setting, for whom a cytology procedure is performed. Cervical samples must be obtainable directly during the consultation at clinical centers with prior Ethics Committee approval. Only participants who meet all inclusion criteria and none of the exclusion criteria will be enrolled
  Interventions: Device: Cytology

INTERVENTIONS:
Device: Cytology — Two cervical samples are collected using a cervical brush or swab, following the standard procedure for cervical cytology. Cells are taken from the cervix using a brush/spatula during a gynecological exam. (1) The first sample is kept in the clinical center's pathology department for examination. (2) The second sample is sent to MiMARK's facilities for the investigational project, where it will be processed and stored for future cohort selection and analysis.

SUMMARY:
CYTOMARK, a non-invasive in vitro diagnostic (IVD) test measuring a defined panel of protein biomarkers in cervical fluid, can accurately detect endometrial cancer in both symptomatic and asymptomatic women at high risk for the disease. The aim of the study consists in validating CYTOMARK's ELISA test, creating and freezing an algorithm detect EC in post-menopausal women with abnormal uterine bleeding (AUB).

ELIGIBILITY:
Inclusion Criteria:

* 1 - Post-menopausal women (≥1 year without menstruation) with AUB who present with: Endometrium > 3mm by transvaginal ultrasound, OR

Endometrium ≤ 3mm who meet at least one of the following criteria:

Persistent symptoms (more than one episode of metrorrhagia) Heterogenous endometrium on transvaginal ultrasonography Risk factors (BMI ≥ 30, use of tamoxifen, hormone replacement therapy (HRT), Lynch syndrome, BRCA mutation.

- 2 - Obtaining written informed consent

Exclusion Criteria:

* 1 - Women with an active pelvic infection. 2 - Women who have had viral infections with evidence of active and latent disease such as Hepatitis B, Hepatitis C, and HIV infection. Patients who have had Hepatitis C in the past but who have been successfully treated and in whom viral replication has not been observed in the last year will be included.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible participants are postmenopausal women presenting with abnormal uterine bleeding (AUB) in a clinical consultation or primary care setting, for whom a cytology procedure is performed. Cervical samples must be obtainable directly during the consultation at clinical centers with prior Ethics Committee approval. Only participants who meet all inclusion criteria and none of the exclusion criteria will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Regulatory Requirements Study | 12 months
  Ensure the stability of the samples under defined conditions (pre-analytica) and the analytical validation of the developed ScreeEC's ELISA test.
Algorithm training with Proprietary Antibodies | 12 months
  Train the current ScreenEC's algorithms defined in MS by assessing the clinical performance of different EC biomarkers individually and in combination detect EC in post- menopausal women with AUB using MiMARK's proprietary antibodies.
Algorithm testing and freeze | 12 months
  To test and freeze the defined algorithm measured with MiMARK's antibodies to rule out EC in post-menopausal women with AUB.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Gil-Moreno, MD, PhD, Principal Investigator — Hospital Universitari Campus Vall d'Hebron
Locations (2):
- Spain (2):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitari Campus Vall d'Hebron, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided